CLINICAL TRIAL: NCT01545531
Title: Two-Point Measurement of Glomerular Filtration Rate by Iohexol Plasma Disappearance
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 6726
Record Dates: First submitted 2011-09-26; First posted 2012-03-06 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Renal Disease; Renal Insufficiency
Keywords: glomerular filtration rate; iohexol; hematopoietic cell transplant; kidney function; gold standard measure; cystatin C.
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for iohexol level, serum creatinine, cystatin C, and hematocrit at baseline, prior to iohexol infusion, 2 hours and 5 hours post iohexol infusion.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Iohexol GFR
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Iohexol, a non-ionic, low osmolar, X-ray contrast medium (OmnipaqueR) that is safe and non-toxic and used for angiographic and urographic procedures, is eliminated from plasma exclusively by glomerular filtration [13]. Study subject will receive 5 ml of iohexol solution (Omnipaque 300, corresponding to 647 mg iohexol per ml or 300 mg iodine per ml) through peripheral IV or central Line infusion over 1-2 minutes followed by 10 ml of saline solution at baseline, day 100 and 1 year after HCT.

SUMMARY:
The purpose of this study is to measure glomerular filtration rate (GFR) by iohexol plasma disappearance (gold standard) and measure serum Cystatin C levels (surrogate marker) in patients enrolled in our prospective study at baseline, day 100 and 1 year after hematopoietic cell transplant and determine if these levels correlate with serum creatinine and an estimated GFR using the Modification of Diet in Renal Disease (MDRD) equation and Schwartz formula in children.

DETAILED DESCRIPTION:
Serum creatinine does not accurately measure kidney function in patients with mild renal insufficiency or in certain other patient populations (for example, individuals with malnutrition, muscle wasting, cancer, or the elderly) [8, 9]. The serum creatinine level and related estimating equations, routinely used clinical measures to estimate kidney function, are dependent on muscle mass, and influenced by age, race, gender, and weight.[10, 11]. Patients undergoing hematopoietic cell transplant may have large fluctuations in their nutritional status, muscle mass and weight that will influence glomerular filtration rates based on estimation equations or serum creatinine levels. In fact, a recently published position paper recommends that research be done specifically to evaluate the accuracy of golemular filtration rate estimating equations in cancer patients "with a particular focus on reducing the influence of confounding factors such as muscle wasting, malnutrition and extracellular fluid volume expansion [12]." Cystatin C is a cysteine protease inhibitor that is expressed by all nucleated cells and is freely filtered by the glomerulus. Serum Cystatin C correlates well with measured glomerular filtration rate and more accurately measures kidney function than does serum creatinine in the elderly, cancer patients, diabetics and renal transplant recipients[9, 13-15]. It is also linearly associated with all cause mortality, cardiovascular mortality and heart failure risk[16]. The gold standard measurements of Golemular filtration rate using inulin or radioisotope-labeled or nonlabeled trace quantities of EDTA, technetium-99-diethylenetriamine pentaacetic acid, iothalamate or iohexol are expensive and time intensive which limits their clinical usefulness. Although the studies done using cystatin C in patients with cancer have reported some conflicting results when comparing cystatin C to estimated GFR measurements, they have generally found it to perform better than serum creatinine [14, 17-20]. Only one study has been done in the HC population to evaluate cystatin C as a measure of renal function and the authors did not include a gold standard measurement for GFR for comparison with cystatin C levels [20]. The authors found elevations in cystatin C in patients after HCT compared to the control group. However, these elevations did not correlate with serum creatinine or creatinine clearance. A plausible conclusion is that serum cystatin C is a more sensitive marker of renal function than the other measures they employed. These authors also did not look at area under the curve, receiver operator characteristic curves or 1/cystatin C curves all of which have been shown to be more accurate and to correlate better with other measures of GFR[21]. Moreover, no long-term studies have been done in this patient population using cystatin C to assess renal function or to define CKD prevalence.

Iohexol, a non-ionic, low osmolar, X-ray contrast medium (OmnipaqueR) that is safe and non-toxic and used for angiographic and urographic procedures, is eliminated from plasma exclusively by glomerular filtration[13]. Iohexol has a molecular weight of 821 daltons, a plasma elimination half-time of ~90 min, is distributed into the extracellular space and has less than 2% plasma protein binding [13, 17]. Iohexol is excreted completely unmetabolized in the urine with 100% recovery within 24 hours after injection [14]. Since iohexol can be quantified in small samples, capillary, as well as venous, sampling can be employed [15]. Extrarenal elimination of iohexol in a setting of reduced GFR is negligible[16]. Iohexol is measured in deproteinized plasma or serum by HPLC. The commercially available preparations contain two isomers of iohexol, both of which are handled similarly by the body [15, 18].

An accurate measure of kidney function is important for clinical management of medications, choice of conditioning regimen, prognosis, and study of treatment toxicities. Establishment of the precise prevalence is needed to design clinical intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* age > 2 years
* follow-up at Seattle cancer care alliance

Exclusion Criteria:

* age <2 years
* history of diabetes mellitus
* inability to return to the SCCA for follow-up at 1 year
* allergy to iodine

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing hematopoietic cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2008-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate | Change from baseline in glomeular filtration rate at different time points after hematopoietic cell transplant
Glomerular Filtration Rate (GFR) | Change from Baseline in GFR at 80 to 100 days post transplant
Glomerular Filtration Rate (GFR) | Change from Baseline in GFR at 1 year post tranplant

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta R. Hingorani, MD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] Beddhu S, Samore MH, Roberts MS, Stoddard GJ, Pappas LM, Cheung AK. Creatinine production, nutrition, and glomerular filtration rate estimation. J Am Soc Nephrol. 2003 Apr;14(4):1000-5. doi: 10.1097/01.asn.0000057856.88335.dd. PMID 12660334
- [Background] Ross EA, Wilkinson A, Hawkins RA, Danovitch GM. The plasma creatinine concentration is not an accurate reflection of the glomerular filtration rate in stable renal transplant patients receiving cyclosporine. Am J Kidney Dis. 1987 Aug;10(2):113-7. doi: 10.1016/s0272-6386(87)80042-2. PMID 3300293
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Fliser D, Franek E, Joest M, Block S, Mutschler E, Ritz E. Renal function in the elderly: impact of hypertension and cardiac function. Kidney Int. 1997 Apr;51(4):1196-204. doi: 10.1038/ki.1997.163. PMID 9083286
- [Background] Levey AS, Atkins R, Coresh J, Cohen EP, Collins AJ, Eckardt KU, Nahas ME, Jaber BL, Jadoul M, Levin A, Powe NR, Rossert J, Wheeler DC, Lameire N, Eknoyan G. Chronic kidney disease as a global public health problem: approaches and initiatives - a position statement from Kidney Disease Improving Global Outcomes. Kidney Int. 2007 Aug;72(3):247-59. doi: 10.1038/sj.ki.5002343. Epub 2007 Jun 13. PMID 17568785
- [Background] Dharnidharka VR, Kwon C, Stevens G. Serum cystatin C is superior to serum creatinine as a marker of kidney function: a meta-analysis. Am J Kidney Dis. 2002 Aug;40(2):221-6. doi: 10.1053/ajkd.2002.34487. PMID 12148093
- [Background] Seronie-Vivien S, Toullec S, Malard L, Thomas F, Durrand V, Chatelut E. Contribution of the MDRD equation and of cystatin C for renal function estimates in cancer patients. Med Oncol. 2006;23(1):63-73. doi: 10.1385/MO:23:1:63. PMID 16645231
- [Background] Visvardis G, Griveas I, Zilidou R, Papadopoulou D, Mitsopoulos E, Kyriklidou P, Manou E, Ginikopoulou E, Meimaridou D, Pavlitou A, Sakellariou G. Glomerular filtration rate estimation in renal transplant patients based on serum cystatin-C levels: comparison with other markers of glomerular filtration rate. Transplant Proc. 2004 Jul-Aug;36(6):1757-9. doi: 10.1016/j.transproceed.2004.06.009. PMID 15350470
- [Background] Shlipak MG, Sarnak MJ, Katz R, Fried LF, Seliger SL, Newman AB, Siscovick DS, Stehman-Breen C. Cystatin C and the risk of death and cardiovascular events among elderly persons. N Engl J Med. 2005 May 19;352(20):2049-60. doi: 10.1056/NEJMoa043161. PMID 15901858
- [Background] Al-Tonbary YA, Hammad AM, Zaghloul HM, El-Sayed HE, Abu-Hashem E. Pretreatment cystatin C in children with malignancy: can it predict chemotherapy-induced glomerular filtration rate reduction during the induction phase? J Pediatr Hematol Oncol. 2004 Jun;26(6):336-41. doi: 10.1097/00043426-200406000-00002. PMID 15167345
- [Background] Holweger K, Bokemeyer C, Lipp HP. Accurate measurement of individual glomerular filtration rate in cancer patients: an ongoing challenge. J Cancer Res Clin Oncol. 2005 Sep;131(9):559-67. doi: 10.1007/s00432-005-0679-7. Epub 2005 Oct 20. PMID 16012866
- [Background] Kleber M, Cybulla M, Bauchmuller K, Ihorst G, Koch B, Engelhardt M. Monitoring of renal function in cancer patients: an ongoing challenge for clinical practice. Ann Oncol. 2007 May;18(5):950-8. doi: 10.1093/annonc/mdm055. Epub 2007 Mar 9. PMID 17351260
- [Background] Demirtas S, Akan O, Can M, Elmali E, Akan H. Cystatin C can be affected by nonrenal factors: a preliminary study on leukemia. Clin Biochem. 2006 Feb;39(2):115-8. doi: 10.1016/j.clinbiochem.2005.10.009. Epub 2005 Dec 6. PMID 16337174
- [Background] Perkins BA, Nelson RG, Ostrander BE, Blouch KL, Krolewski AS, Myers BD, Warram JH. Detection of renal function decline in patients with diabetes and normal or elevated GFR by serial measurements of serum cystatin C concentration: results of a 4-year follow-up study. J Am Soc Nephrol. 2005 May;16(5):1404-12. doi: 10.1681/ASN.2004100854. Epub 2005 Mar 23. PMID 15788478